CLINICAL TRIAL: NCT01882660
Title: Pre-operative Decitabine in Colon Cancer: a Proof of Principle Study
Acronym: DECO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusion of patients was slow. Could not reach the target within the studyperiod.
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, H.W.M. van Laarhoven, Dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NL44048.018.13
Record Dates: First submitted 2013-05-24; First posted 2013-06-20 (Estimated); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Decitabine treatment (Experimental): Treatment with decitabine
  Interventions: Drug: Decitabine

INTERVENTIONS:
Drug: Decitabine

SUMMARY:
Background of the study: Colon cancer is the second leading cause of cancer-related death world wide.

Although patients presenting with early disease (stage I-III) can be cured, prognosis varies from 90% in stage I to 50-80% in stage II and III. Therefore, prevention of metastases after early disease is of utmost importance. Derepression of Wnt targets may provide a novel target for therapy.

Objectives: The primary objective of the study is to assess in patients with primary colon cancer whether short-course pre-operative treatment with decitabine can increase Wnt target gene expression as measured in resected tumors compared to pretreatment biopsies. The secondary objective of the study is to assess in patients with primary colon cancer whether short-course pre-operative treatment with decitabine can revert CpG methylation and induce more favorable tumor characteristics as measured in resected tumors compared to pretreatment biopsies. The tertiary objective is to compare changes in Wnt target gene expression, CpG methylation and tumor characteristics for Wnt methylated and nonmethylated tumors as measured in resected tumors compared to pretreatment biopsies and identify new stratification markers.

DETAILED DESCRIPTION:
Rationale: Colon cancer is the second leading cause of cancer-related death world wide.

Although patients presenting with early disease (stage I-III) can be cured, prognosis varies from 90% in stage I to 50-80% in stage II and III. Therefore, prevention of metastases after early disease is of utmost importance. Extensive studies of the Wnt signal cascade have elucidated its role in colorectal cancer development and proliferation. Several well-known targets of the Wnt-cascade, like DKK1, APCDD1 and AXIN2, serve as feedback inhibitors and likely prevent pathway hyperactivation. Therefore, loss of these control mechanisms, for example due to repression of Wnt targets by CpG island methylation, serves as a potent proliferative signal. Recently, we identified a subset of colon cancers that are typified by CpG island methylation of specific Wnt target genes and have a poor prognosis. Moreover, in preclinical studies we showed that derepression of Wnt-targets by the demethylating agent decitabine resulted in tumor growth suppression. Thus, derepression of Wnt targets may provide a novel target for therapy. Objectives: The primary objective of the study is to assess in patients with primary colon cancer whether short-course pre-operative treatment with decitabine can increase Wnt target gene expression as measured in resected tumors compared to pretreatment biopsies. The secondary objective of the study is to assess in patients with primary colon cancer whether short-course pre-operative treatment with decitabine can revert CpG methylation and induce more favorable tumor characteristics as measured in resected tumors compared to pretreatment biopsies. The tertiary objective is to compare changes in Wnt target gene expression, CpG methylation and tumor characteristics for Wnt methylated and nonmethylated tumors as measured in resected tumors compared to pretreatment biopsies and identify new stratification markers.

Study design: Interventional study.

Study population:

Patients > 18 yr old with histopathologically proven or high suspicion of colon cancer.

Intervention: In patients with proven colon cancer, five extra biopsies will be taken from the tumour during endoscopy to determine CpG methylation of Wnt target genes in fresh tumor samples. Next, these patients will pre-operatively receive decitabine as a single intravenous infusion at a dose of 45 mg/m2 over 6 hr. After resection, Wnt target gene expression and CpG methylation of Wnt target genes will again be determined in fresh tumor samples.

Main study parameters: The primary study parameter is Wnt target gene expression (APCDD1, AXIN2, DKK1, LGR5 and ASCL2). Secondary study parameters are Wnt target and CIMP gene methylation, beta-catenin localization, proliferation (Ki-67), apoptosis (TUNEL and M30 assay) and tumor differentiation.

ELIGIBILITY:
In- and exclusion criteria first part:

In order to participate in the first part of the study, five extra fresh biopsies to determine tumor methylation status, a subject must meet all of the following criteria:

Inclusion criteria:

1. Biopsy proven colon cancer or high suspicion of colon cancer on a previous endoscopy.
2. Planned endoscopy.
3. Age ≥ 18yr.
4. ECOG/ WHO performance 0-2.
5. Written informed consent.

Exclusion criteria:

1. Any psychological, familial, sociological or geographical condition potentially hampering adequate informed consent or compliance with the study protocol.

In- and exclusion criteria second part:

In order to participate in the second part of the study - treatment with decitabine - a subject must meet all of the following criteria:

Inclusion criteriä:

1. Patients with biopsy proven colon cancer who will undergo primary tumor resection.
2. Age ≥ 18yr.
3. ECOG/ WHO performance 0-2.
4. Adequate bone marrow function (ANC>1500/mm3, hemoglobin>9g/dL (which may be obtained by transfusions), platelets>100,000)
5. Adequate hepatic function (AST and ALT <2.5x upper limit of normal (ULN)).
6. Adequate renal function (Serum creatinine ≤1.5 x ULN or calculated creatinine of >50ml/min)
7. Women of child-bearing age must be willing to use adequate contraception and have negative serum or urine pregnancy test within 3 days prior to registration.
8. Written informed consent.

Exclusion criteria:

1. Known hypersensitivity to decitabine or its additives.
2. Surgery not planned according to time frame of the study,
3. Other systemic or local treatment of the primary tumor in the waiting time until surgery.
4. Administration of any experimental drug within 60 days prior to the first dose of decitabine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-07; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Wnt target gene expression (APCDD1, AXIN2, DKK1, LGR5 and ASCL2) | 30 minutes after surgery
  The primary objective of the study is to assess whether short-course pre-operative treatment with the demethylating agent decitabine can increase Wnt target gene expression as measured in resected tumors compared to pretreatment biopsies in patients with primary colon cancer.

SECONDARY OUTCOMES:
Wnt target methylation. | 30 minutes after surgery
  The secondary objective of the study is to assess whether short-course pre-operative treatment with decitabine can revert CpG methylation and induce more favorable tumor characteristics as measured in resected tumors compared to pretreatment biopsies in patients with primary colon cancer.
CIMP gene methylation | 30 minutes after surgery
  See above
Beta-catenin localisation | 30 minutes after surgery
  See above
Proliferation (Ki-67) | 30 minutes after surgery
  See above
Apoptose (TNEL en M30 assay) | 30 minutes after surgery
  See above.
Tumor differentiation | 30 minutes after surgery
  See above

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands